CLINICAL TRIAL: NCT00192114
Title: A Phase 2 Study of Oral Enzastaurin HCl in Patients With Metastatic Colorectal Cancer
Brief Title: Enzastaurin for Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9098; H6Q-MC-JCAR (Other: Eli Lilly and Company)
Record Dates: First submitted 2005-09-14; First posted 2005-09-19 (Estimated); Results first posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-07

CONDITIONS: Colonic Neoplasms
MeSH Terms: conditions — Colonic Neoplasms | interventions — enzastaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enzastaurin HCl (Experimental)
  Interventions: Drug: Enzastaurin HCl

INTERVENTIONS:
Drug: Enzastaurin HCl — 1200 milligrams (mg) loading dose orally, then 500 mg, orally, daily, up to six 28-day cycles.
  Other Names: LY317615

SUMMARY:
Enzastaurin given daily to participants with colorectal cancer who have Stage 4 disease and have not received prior chemotherapy for advanced colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with colorectal cancer that is advanced or metastatic (has spread to other parts of the body); able to visit the doctor's office every 28 days for at least 6 months; able to swallow tablets

Exclusion Criteria:

* women cannot be pregnant or breastfeeding; no history of significant heart disease or any other significant medical problems as determined by the participant's physician

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2005-08; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- Denmark (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Odense
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vejle
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Uppsala, Sweden

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participant flow reports those who discontinued from study drug.
Groups:
- Enzastaurin HCl: 1200 milligrams (mg) administered orally as a loading dose then 500 mg administered orally, once daily, for up to six 28-day cycles.
Period: Overall Study
Arm/Group | Enzastaurin HCl
Started | 28
Received at Least 1 Dose of Study Drug | 28
Completed | 4
Not Completed | 24
Not completed — Objective Tumor Progression | 19
Not completed — Adverse Event | 2
Not completed — Clinical Progression | 2
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Enzastaurin HCl: 1200 milligrams (mg) administered orally as a loading dose, then 500 mg administered orally, once daily, for up to six 28-day cycles.
Arm/Group | Enzastaurin HCl
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.75 (8.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Denmark | 13
  Sweden | 15
Eastern Cooperative Oncology Group (ECOG) [Count of Participants; unit: Participants] — ECOG performance status:
  0 - Fully active, able to carry on all pre-disease performance without restriction.
  1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, for example, light house work, office work.
  Participants
    0 | 24
    1 | 4
Pathological Diagnosis [Count of Participants; unit: Participants] — Pathological diagnosis at baseline.
  Participants
    Adenocarcinoma colon | 16
    Adenocarcinoma rectum | 10
    Colorectal Cancer | 1
    Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression Free Survival (PFS) at 6 Months
Description: PFS defined as time from date of first dose of enzastaurin to first date of documented progressive disease (PD) or date of death (any cause), whichever occurred first. Using Response Evaluation Criteria in Solid Tumors (RECIST v1.0) PD defined as ≥20% increase in sum of the longest diameter (LD) of target lesions, taking as reference smallest sum LD recorded since treatment started or appearance of ≥1 new lesions. Participants not known to have died as of data-inclusion cut-off date and who did not have PD, PFS was censored at date of last progression-free disease assessment prior to date of any post discontinuation anticancer therapy. Participants who took any subsequent systemic anticancer therapy prior to PD or death, PFS was censored at date of last progression-free disease assessment prior to the date of any post discontinuation anticancer therapy. PFS at 6 months = participants who were progression free and alive at 6 months divided by the number of treated participants x 100.
Time Frame: Baseline to 6 months
Population: All randomized participants who received at least 1 dose of study drug. Censored participants =5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzastaurin HCl
Number analyzed (Participants) | 28
percentage of participants | 27.50 [12.53 to 44.82]

2. Secondary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR) [Objective Response Rate (ORR)]
Description: Objective response rate during treatment was defined as the number of participants with documented complete response (CR) or partial response (PR) divided by the total number of participants. CR and PR defined using Response Evaluation Criteria in Solid Tumors (RECIST v1.0). CR defined as the disappearance of all target and non-target lesions and normalization of tumor marker levels in non-target lesions. PR defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Percentage of participants with CR or PR (ORR) was the number of participants with documented CR or PR divided by the total number of treated participants x 100.
Time Frame: Baseline to measured progressive disease (PD) up to 24 months
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzastaurin HCl
Number analyzed (Participants) | 28
percentage of participants | 0 [NA to NA] — Not evaluable, no participants achieved CR or PR.

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of the first dose of enzastaurin to the date of death from any cause. Survival time was censored at the date of the last contact for participants who were still alive.
Time Frame: Baseline to date of death from any cause up to 24 months
Population: All randomized participants who received at least 1 dose of study drug. Censored participants =23.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzastaurin HCl
Number analyzed (Participants) | 28
months | 23.38 [NA to NA] — Only 5 of 28 participants had events observed. Due to the high censoring rate and due to the pattern of censoring, the median is estimable but the 95% CI is undefined.

4. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of the first dose of enzastaurin to the first date of documented progressive disease (PD) or the date of death from any cause, whichever occurred first. Participants who were not known to have died as of the data-inclusion cut-off date, and who did not have PD, PFS was censored at the date of the last progression-free disease assessment date prior to the date of any post discontinuation anticancer therapy. Participants who took any subsequent systemic anticancer therapy prior to PD or death, PFS was censored at the date of the last progression-free disease assessment prior to the date of any post discontinuation anticancer therapy.
Time Frame: Baseline to measured PD up to 9 months
Population: All randomized participants who received at least 1 dose of study drug. Censored participants =5.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzastaurin HCl
Number analyzed (Participants) | 28
months | 1.89 [1.77 to 4.52]

5. Secondary Outcome: Duration of Stable Disease (SD)
Description: Duration of SD measured from date of first dose of enzastaurin to date of documented progressive disease (PD) or date of death from any cause, whichever occurred first, using Response Evaluation Criteria in Solid Tumors (RECIST v1.0). PD was defined as ≥20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD since treatment began or appearance of ≥1 new lesions. SD was defined as no improvement and not meeting the requirements of PD using smallest sum LD since treatment began as reference. Participants with SD (or better) who had not died at data-inclusion cut-off date without PD, or participants who took subsequent systemic anticancer therapy prior to PD or death, duration was censored at date of last progression-free disease assessment prior to the date of post discontinuation anticancer therapy.
Time Frame: Time from SD to measured PD up to 9 months
Population: Subset of all randomized participants who received at least 1 dose of study drug who achieved complete response (CR), partial response (PR) or SD. Censored participants =5.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzastaurin HCl
Number analyzed (Participants) | 12
months | 6.13 [3.64 to NA] — Too few observations to determine upper level of 95% confidence interval.

6. Secondary Outcome: Time to Treatment Response
Description: Time to treatment response was defined as date of first dose of study drug to the date of confirmed complete response (CR) or partial response (PR) using Response evaluation Criteria in Solid Tumors (RECIST v1.0) criteria. CR was defined as the disappearance of all target and non-target lesions and normalization of tumor marker levels in non-target lesions. PR was defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Time to treatment response was not evaluable, as there were no participants with CR or PR.
Time Frame: Baseline to date of confirmed response up to 24 months
Population: Zero participants were analyzed.
Arm/Group | Enzastaurin HCl
Number analyzed (Participants) | 0

7. Secondary Outcome: Duration of Complete Response (CR) or Partial Response (PR) (Duration of Response)
Description: The duration CR or PR was defined as the time from first objective status assessment of CR or PR to the first date of documented progressive disease (PD) or death from any cause. CR and PR were determined using Response evaluation Criteria in Solid Tumors (RECIST v1.0) criteria. CR was defined as the disappearance of all target and non-target lesions and normalization of tumor marker levels in non-target lesions. PR was defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. PD defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of 1 or more new lesions. Duration of response was not evaluable, as there were no participants with CR or PR.
Time Frame: Time from response to PD
Population: Zero participants were analyzed.
Arm/Group | Enzastaurin HCl
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Participants With Adverse Events (AEs) or Who Died
Description: Clinically significant events were defined as serious AEs (SAEs) and other non-serious AEs (regardless of causality). A summary of SAEs and other non-serious adverse events (AEs) regardless of causality is located in the Reported Adverse Events module. The number of participants who died included those who died due to an SAE (any cause) while on study and those who died due to progressive disease (PD) during the 30-day post-study discontinuation follow-up.
Time Frame: Baseline to study completion up to 24 months and 30-day post-study discontinuation
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzastaurin HCl
Number analyzed (Participants) | 28
Participants
  Serious AEs | 4
  AEs | 22
  Died due to PD during 30-day follow-up | 2
  Died due to SAE while on study | 1

9. Secondary Outcome: Change From Baseline in QTc Interval
Description: QTc interval was a measure of time between the start of the Q wave and the end of the T wave and is dependent on the heart rate. A QTc interval adjusted using Bazette's correction (QTcB) was used in order to aid interpretation.
Time Frame: Baseline, Cycle 1 Day 1 and Cycle 2 Day 1 of 28-day cycles
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Arm/Group | Enzastaurin HCl
Number analyzed (Participants) | 28
milliseconds (msec)
  Cycle 1 Day 1 | 2.07 (16.21)
  Cycle 2 Day 1 | 7.30 (15.76)

10. Secondary Outcome: Pharmacokinetics-Minimum Observed Concentration (Cmin) of Total Analytes
Description: Cmin of enzastaurin + LSN326020 (a metabolite of LY317615) after loading dose in Cycle 1 and at a steady state during Cycles 2 and 3.
Time Frame: Cycle 1 Day 2-predose, Cycle 2 Day 1-predose and Cycle 3 Day 1-predose of 28-day cycles
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: nanomoles per liter (nmol/L)
Arm/Group | Enzastaurin HCl
Number analyzed (Participants) | 28
nanomoles per liter (nmol/L)
  Cycle 1 Day 2 | 2180 (1343)
  Cycle 2 Day 1: number analyzed (Participants) | 19
  Cycle 2 Day 1 | 1723 (2042)
  Cycle 3 Day 1: number analyzed (Participants) | 10
  Cycle 3 Day 1 | 1374 (936)

11. Secondary Outcome: Change From Baseline in Carcinoembryonic Antigen (CEA) Response at Each Cycle
Description: CEA levels were measured to detect potentially rapid-growing tumors in participants who received enzastaurin.
Time Frame: Baseline and Cycles 1, 2, 3, 4, 5, 6 (28-day cycles)
Population: All participants with both baseline and post baseline CEA measurements.
Measure: Median (Inter-Quartile Range); unit: micrograms per liter (mcg/L)
Arm/Group | Enzastaurin HCl
Number analyzed (Participants) | 27
micrograms per liter (mcg/L)
  Cycle 1: number analyzed (Participants) | 10
  Cycle 1 | 0.20 [0.00 to 0.70]
  Cycle 2: number analyzed (Participants) | 19
  Cycle 2 | 0.30 [-1.60 to 36.60]
  Cycle 3: number analyzed (Participants) | 14
  Cycle 3 | 0.90 [0.10 to 2.30]
  Cycle 4: number analyzed (Participants) | 9
  Cycle 4 | 0.80 [0.40 to 3.30]
  Cycle 5: number analyzed (Participants) | 8
  Cycle 5 | 0.80 [0.35 to 3.40]
  Cycle 6: number analyzed (Participants) | 4
  Cycle 6 | 0.35 [-0.25 to 14.85]

12. Other Pre Specified Outcome: Change From Baseline in Vascular Endothelial Growth Factor (VEGF) to Cycle 2 and Cycle 3
Description: VEGF levels were measured to detect potentially rapid-growing tumors in participants who received enzastaurin.
Time Frame: Baseline, Cycle 2 and Cycle 3 (28-day cycles)
Population: Participants with both baseline and post-baseline VEGF measurements.
Measure: Median (Inter-Quartile Range); unit: picograms per liter (pg/L)
Arm/Group | Enzastaurin HCl
Number analyzed (Participants) | 28
picograms per liter (pg/L)
  Cycle 2: number analyzed (Participants) | 7
  Cycle 2 | 0.50 [-4.40 to 34.30]
  Cycle 3: number analyzed (Participants) | 4
  Cycle 3 | -0.10 [-2.40 to 3.15]

ADVERSE EVENTS:
Description: Study-specific clinical outcomes due to progressive disease were not considered to be a serious adverse event (SAE) unless the investigator deemed it related to the use of the study drug.
Groups:
- Enzastaurin HCl: 1200 milligrams (mg) of enzastaurin HCl administered orally as a loading dose then 500 mg, administered orally once daily up to six 28-day cycles.
Arm/Group | Enzastaurin HCl
Serious Adverse Events (participants affected / at risk) | 4/28
Other Adverse Events (participants affected / at risk) | 22/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzastaurin HCl (N=28)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzastaurin HCl (N=28)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Faeces discoloured (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 6 (6)
Vomiting (Gastrointestinal disorders) | 2 (2)
Chills (General disorders) | 2 (2)
Fatigue (General disorders) | 7 (7)
Nasopharyngitis (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2)
Blood creatinine increased (Investigations) | 2 (2)
Blood urea (Investigations) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3)
Chromaturia (Renal and urinary disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days